CLINICAL TRIAL: NCT06861621
Title: STRucturation of Transcript Analysis of Genes Involved in Hereditary Cancers in Normandy and Hauts de France
Brief Title: STRucturation of Transcript Analysis of Genes Involved in Hereditary Cancers
Acronym: STRATEGIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/310/OB; IDRCB : 2023-A00488-37 (Other: ANSM)
Record Dates: First submitted 2025-02-19; First posted 2025-03-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: hereditary predisposition to cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An analysis of the predisposition genes will be carried out on the patients' DNA as part of the treatment after informed consent has been obtained. If patients do not object to taking part in the STRATEGIC study, an additional blood sample (PAXEGENE tube for RNA) will be taken during the blood test as part of the treatment. The major predisposing genes, breast/ovarian and digestive, will then be studied using both DNA and RNA. The results will be analysed centrally and used to evaluate this new diagnostic strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Molecular diagnosis using high throughput sequencing has become an essential part of oncogenetic care, making it possible to identify people at risk, to guide surveillance, and to direct preventive surgery and treatment. The quality of this 'precision' care depends on the quality of the interpretation of the genomic variants identified. To be usable in oncogenetics, a genomic variant must be correctly interpreted: pathogenic, benign or of uncertain significance (VSI). The impact of these DNA variants (VSI) on RNA is particularly important for interpretation. Today, due to a lack of resources, joint and systematic DNA/RNA analysis is never carried out. This has inevitably meant that a number of situations of interest have been overlooked. It is now important to go a step further and organise a visible and reliable circuit, allowing routine access to these studies for patients.

DETAILED DESCRIPTION:
Systematic DNA/RNA analysis is never carried out using the current approach, due to a lack of resources. Strategies recommend pre-screening variants using in silico analysis, followed by RNA studies targeting variants of interest.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patients seen in oncogenetic consultations and who have given their informed consent for genetic analysis in the context of a major predisposition to breast, ovarian or digestive cancer.
* Person who has read and understood the information note and does not object to taking part in the study
* Membership of a social security scheme

Exclusion Criteria:

* Minors
* Persons deprived of their liberty or adults under guardianship or incapable of giving their consent
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive people seen in oncogenetic consultations for a hereditary predisposition to breast, ovarian or digestive cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Relevance of a joint systematic DNA/RNA study | Baseline
  The main objective is to assess the relevance of a joint, systematic DNA/RNA study when managing patients in oncogenetic consultations, without any pre-requisites based on personal or family history criteria or on in silico predictions of a DNA variant. The study compares the diagnostic yield (Diagnostic yield corresponds to the rate of patients with a positive molecular diagnosis, confirming a hereditary predisposition to cancer, as a proportion of all patients analysed) obtained using the current approach (DNA alone, then possible use of RNA analyses in rare cases) and that obtained in this study (DNA and RNA systematically).

SECONDARY OUTCOMES:
Structuring the transcript analysis circuit | 6 months
  Structuring the transcript analysis circuit to ensure that results are compatible with the clinical management of patients. The study is designed to compare the mutational yield between the current strategy and that proposed by the study

CONTACTS AND LOCATIONS:
Overall Officials: Claude HOUDAYER, Professor, Principal Investigator — Molecular Genetics Department, UH of Rouen
Locations (2):
- France (2):
  - Service Oncogénétique Centre François Baclesse, Caen
  - Clinique de génétique médicale Guy Fontaine de l'hopital de Flandre CHRU de Lille, Lille

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.